CLINICAL TRIAL: NCT02311244
Title: The Sapienza University Mortality and Morbidity Events Rate (SUMMER) Study in Diabetes: Identification of New Molecular Promoters of Mortality and Morbidity in Patients With Type 2 Diabetes Mellitus
Brief Title: The Sapienza University Mortality and Morbidity Events Rate (SUMMER) Study in Diabetes
Acronym: SUMMER
Status: Completed | Type: Observational
Sponsor: University of Roma La Sapienza (Other)
Collaborators: Campus Bio-Medico University (Other); Ospedale Sandro Pertini, Roma (Other); Azienda Ospedaliera San Camillo Forlanini (Other); University of Cagliari (Other); Casa Sollievo della Sofferenza IRCCS (Other)
Responsible Party: Principal Investigator, Vincenzo Trischitta, MD, Professor of Endocrinology, University of Roma La Sapienza
Other Study IDs: URomLS-01-2014
Record Dates: First submitted 2014-11-24; First posted 2014-12-08 (Estimated); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: All-cause mortality; Cardiovascular mortality; Myocardial infarction; Stroke; Dialysis
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Myocardial Infarction; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum and urine
Oversight: Data Monitoring Committee: No

SUMMARY:
This observational study is aimed at identifying new molecular promoters of mortality (and morbidity) in patients with type 2 diabetes mellitus (T2DM).

DETAILED DESCRIPTION:
Background Mortality rate of diabetic patients is about twice as much that of non-diabetic individuals of similar age; this makes diabetes a leading risk factor for mortality, especially of cardiovascular origin, which accounts for 2.9 million global events yearly. Such scenario is expected to further deteriorate, given that the prevalence of type 2 diabetes mellitus (T2DM), by far the most common form of diabetes comprising more than 90% of all diabetic individuals, is increasing worldwide. Predicting such devastating event is, therefore, urgently needed in order to target aggressive prevention strategies in high risk T2DM patients.

Aims This observational study is aimed at identifying new molecular promoters of all-cause mortality in patients with T2DM.

Secondary endpoints are to identify in these individuals molecular markers of

* cardiovascular mortality;
* myocardial infarction;
* stroke;
* dialysis.

Other pre-specified endpoints are to assess in these subjects:

* LADA;
* severe hypoglycemic episodes;
* revascularization procedures;
* hospitalization for heart failure;
* other co-morbidities (cancer - at follow-up only, liver disease, chronic obstructive pulmonary disease, autoimmune and endocrine disorders, other - non-diabetic - renal diseases, fractures, cognitive impairment).

Patients A total of 5,000 patients with T2DM of both sexes will be recruited. Measures The following parameters will be recorded as exposure variables at baseline.

* Age, BMI, waist circumference, systolic and diastolic pressure;
* Lifestyle habits, including diet, physical activity (both by validated questionnaires) and smoking.
* Menopausal state (for women).
* Family history of diabetes (3 consecutive generations).
* Family history of cardiovascular disease (first degree relatives).
* Diabetes duration.
* Severe (requiring assistance) hypoglycemic episodes (per year).
* Myocardial infarction, stroke, ulcer/gangrene/amputation, coronary and peripheral revascularization, hospitalization for heart failure, dialysis (at follow-up only).
* Glucose, HbA1c, creatinine, uric acid, total and HDL cholesterol, triglycerides, high sensitive C reactive protein, testosterone, Vitamin D, uric acid levels, white blood cells counting, urinary albumin creatinine ratio (ACR)
* Current glucose-, lipid-, blood pressure-lowering and anti-platelet or anti-coagulant treatment.
* Other relevant treatments (steroids, NSAIDs, immunomodulators, androgens, estrogens, anti-fracturative therapy).
* Main co-morbidities (cancer, chronic liver disease, chronic obstructive pulmonary disease, autoimmune and endocrine disorders, other - non-diabetic - renal diseases, fractures, cognitive impairment).

The following parameters will be assessed at baseline only:

* GADAs (by a radiobinding assay using in vitro translated [35S] methionine-labelled GAD65) and IA-2 antibodies (by radioimmunoprecipitation assays) to identify subjects with LADA.
* Genomic (common and rare variants in genes of interest according to a pathway-centric approach by means of Affymetrix platforms), transcriptomic (differential levels of mRNA by GeneChip Human Gene 1.0 ST Array from Affymetrix) and metabolomic by a combination of ultra-pressure liquid chromatography and gas chromatography coupled to mass spectrometry) analysis.

Measurements of testosterone, Vitamin D, GADAs and IA-2 antibodies as well as gnomic, transcriptomic and metabolomic analysis will be centralized.

Time schedule Recruitment of patients will last approximately 3 years. The enrolled patients will be followed for at least 5 years with yearly visits and telephone calls or consultation of death records in case of drop-out for unknown reasons.

ELIGIBILITY:
Inclusion Criteria:

Type 2 diabetes mellitus

Exclusion Criteria:

* Severe psychiatric illnesses
* End-stage renal disease and dialysis
* Cirrhosis
* Any active cancer

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Secondary care outpatients clinic
Sampling Method: Probability Sample
Enrollment: 5139 (Actual)
Dates: Start 2014-01; Primary Completion 2020-12 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
Number of all-cause deaths | 5 years
  Number of participants who die for all causes and time of occurrence of such events

SECONDARY OUTCOMES:
Number of cardiovascular deaths | 5 years
  Number of participants who die for cardiovascular causes and time of occurrence of such events
Number of subjects with myocardial infarction | 5 years
  Number of participants who develop myocardial infarction and time of occurrence of such events
Number of subjects with stroke | 5 years
  Number of participants who develop stroke and time of occurrence of such events
Number of subjects entering dialysis | 5 years
  Number of participants who enter dialysis and time of occurrence of such events

CONTACTS AND LOCATIONS:
Overall Officials: Vincenzo Trischitta, MD, Principal Investigator — University of Roma La Sapienza; Giuseppe Pugliese, MD, PhD, Study Director — University of Roma La Sapienza
Locations (1):
- University of Roma La Sapienza, Rome, RM, Italy

REFERENCES:
- [Background] Rao Kondapally Seshasai S, Kaptoge S, Thompson A, Di Angelantonio E, Gao P, Sarwar N, Whincup PH, Mukamal KJ, Gillum RF, Holme I, Njolstad I, Fletcher A, Nilsson P, Lewington S, Collins R, Gudnason V, Thompson SG, Sattar N, Selvin E, Hu FB, Danesh J; Emerging Risk Factors Collaboration. Diabetes mellitus, fasting glucose, and risk of cause-specific death. N Engl J Med. 2011 Mar 3;364(9):829-841. doi: 10.1056/NEJMoa1008862. PMID 21366474
- [Background] Roglic G, Unwin N, Bennett PH, Mathers C, Tuomilehto J, Nag S, Connolly V, King H. The burden of mortality attributable to diabetes: realistic estimates for the year 2000. Diabetes Care. 2005 Sep;28(9):2130-5. doi: 10.2337/diacare.28.9.2130. PMID 16123478
- [Background] De Cosmo S, Copetti M, Lamacchia O, Fontana A, Massa M, Morini E, Pacilli A, Fariello S, Palena A, Rauseo A, Viti R, Di Paola R, Menzaghi C, Cignarelli M, Pellegrini F, Trischitta V. Development and validation of a predicting model of all-cause mortality in patients with type 2 diabetes. Diabetes Care. 2013 Sep;36(9):2830-5. doi: 10.2337/dc12-1906. Epub 2013 May 1. PMID 23637348
- [Background] Hong Kong Diabetes Registry; Yang X, So WY, Tong PC, Ma RC, Kong AP, Lam CW, Ho CS, Cockram CS, Ko GT, Chow CC, Wong VC, Chan JC. Development and validation of an all-cause mortality risk score in type 2 diabetes. Arch Intern Med. 2008 Mar 10;168(5):451-7. doi: 10.1001/archinte.168.5.451. PMID 18332288
- [Background] Wells BJ, Jain A, Arrigain S, Yu C, Rosenkrans WA Jr, Kattan MW. Predicting 6-year mortality risk in patients with type 2 diabetes. Diabetes Care. 2008 Dec;31(12):2301-6. doi: 10.2337/dc08-1047. Epub 2008 Sep 22. PMID 18809629
- [Background] McEwen LN, Karter AJ, Waitzfelder BE, Crosson JC, Marrero DG, Mangione CM, Herman WH. Predictors of mortality over 8 years in type 2 diabetic patients: Translating Research Into Action for Diabetes (TRIAD). Diabetes Care. 2012 Jun;35(6):1301-9. doi: 10.2337/dc11-2281. Epub 2012 Mar 19. PMID 22432119
- [Derived] Maddaloni E, Coraggio L, Amendolara R, Baroni MG, Cavallo MG, Copetti M, Cossu E, D'Angelo P, D'Onofrio L, Cosmo S, Leonetti F, Morano S, Morviducci L, Napoli N, Prudente S, Pugliese G, Park K, Holman RR, Trischitta V, Buzzetti R; SUMMER Study in Diabetes Group. Association of osteocalcin, osteoprotegerin, and osteopontin with cardiovascular disease and retinopathy in type 2 diabetes. Diabetes Metab Res Rev. 2023 Jul;39(5):e3632. doi: 10.1002/dmrr.3632. Epub 2023 Mar 20. PMID 36880127
- [Derived] Barchetta I, Capoccia D, Baroni MG, Buzzetti R, Cavallo MG, De Cosmo S, Leonetti F, Leotta S, Morano S, Morviducci L, Prudente S, Pugliese G, Trischitta V; SUMMER Study in Diabetes Group. The "Sapienza University Mortality and Morbidity Event Rate (SUMMER) study in diabetes": Study protocol. Nutr Metab Cardiovasc Dis. 2016 Feb;26(2):103-8. doi: 10.1016/j.numecd.2015.09.009. Epub 2015 Oct 9. PMID 26698225
- See also: Study webpage — http://www.summerstudyindiabetes.it/